CLINICAL TRIAL: NCT06581406
Title: A Randomized, Phase 2/3, Open-Label Study to Investigate the Efficacy and Safety of RP2 in Combination With Nivolumab Versus Ipilimumab in Combination With Nivolumab in Immune Checkpoint Inhibitor-Naïve Adult Patients With Metastatic Uveal Melanoma
Brief Title: A Randomized, Phase 2/3 Study to Investigate the Efficacy and Safety of RP2 in Combination With Nivolumab in Immune Checkpoint Inhibitor-Naïve Adult Patients With Metastatic Uveal Melanoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Replimune Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP2-202
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Uveal Melanoma
Keywords: Metastatic; Uveal; Melanoma; Nivolumab; Ipilimumab; Randomized; Immune checkpoint inhibitor-naïve; RP2; Oncolytic viruses; HSV-1
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis; Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: The study will consist of 3 periods: Screening, Treatment, and Follow-up.
  * 28-day Screening Period
  * Treatment Period: Tumor measurements will be assessed every 12 weeks (Q12W)
  * Safety Follow-Up - up to 100 days after the last dose of study drug.
  * Efficacy Follow-Up,Tumor measurements by serial radiographic imaging Q12W
  * Survival Follow-Up, survival information will be collected every 3 months for a minimum of 3 years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test Arm: RP2 + nivolumab (Experimental): RP2 (Oncolytic virus) and Nivolumab (programmed death receptor-1 (PD-1) inhibitor)
  Interventions: Biological: RP2; Biological: Nivolumab
- Control Arm (Active Comparator): ipilimumab + nivolumab (Experimental): Immune Checkpoint inhibitor combination
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Biological: RP2 — Genetically modified herpes simplex type 1 virus for tumor lysis and immune stimulation.
  Arms: Test Arm: RP2 + nivolumab
Biological: Ipilimumab — Ipilimumab: human cytotoxic T-lymphocyte antigen 4 (CTLA-4)-blocking antibody
  Other Names: Yervoy
  Arms: Control Arm (Active Comparator): ipilimumab + nivolumab
Biological: Nivolumab — Nivolumab: Anti-PD-1 Monoclonal antibody
  Other Names: Opdivo

SUMMARY:
The purpose of this study is to measure the clinical benefits of the combination of RP2 and nivolumab as compared with the combination of nivolumab and ipilimumab in patients with metastatic uveal melanoma who have not been treated with immune checkpoint inhibitor therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients who are 18 years of age or older at the time of signed informed consent.
* Patients with confirmed diagnosis of metastatic Uveal melanoma not amenable to surgical resection.
* Has at least 1 measurable and injectable tumor of ≥ 1 cm in longest diameter (≥ 1.5 cm in the shortest axis for a lymph node [LN]) that is amenable to serial RP2 injections.
* Must be willing to provide tumor biopsy samples.
* LDH ≤ 2 × upper limit of normal (ULN).
* Has adequate hematologic, hepatic and renal function
* Prothrombin time (PT) ≤ 1.5 × ULN (or international normalization ratio [INR] ≤ 1.3) and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
* Life expectancy of > 6 months as estimated by the Investigator.

Key Exclusion Criteria:

* Any exposure to immune checkpoint inhibitor (ICIs) since the time of first being diagnosed with uveal melanoma.
* Known acute or chronic Hepatitis B or C infection or human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
* Current active significant herpetic infections or prior complications of HSV-1 infection.
* Any central nervous system (CNS) involvement of melanoma, including carcinomatous meningitis.
* Major surgery ≤ 2 weeks prior to the first dose of study intervention.
* Any bleeding, thrombotic and/or other event that places the patient at an unacceptable risk of complications of intratumoral therapy.
* Active, known, or suspected autoimmune disease requiring systemic treatment.
* Prior treatment with an oncolytic virus.
* Requires intermittent or chronic use of systemic (oral or IV) antivirals with known antiherpetic activity (eg, acyclovir).
* Systemic anticancer therapy or prior radiotherapy within 2 weeks of the first dose.
* Has received Investigation agent within 4 weeks or 5 half-lives (whichever longer) prior to the first dose.
* Conditions requiring treatment with immunosuppressive doses (> 10 mg per day of prednisone or equivalent) of systemic corticosteroids other than for corticosteroid replacement therapy within 14 days after enrollment.

Additional inclusion/ exclusion criteria are outlined in the study protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From Day 1 up to 3 years after last dose.
  OS is the time from the date of randomization to death from any cause.
Progression Free Survival (PFS) | From Day 1 up to 3 years after last dose.
  PFS is the time from randomization to first evidence of confirmed disease progression as assessed by BICR per RECIST 1.1 or death from any cause.

SECONDARY OUTCOMES:
Number of patients with treatment-emergent adverse events (TEAEs) | From first dose up to 100 days after last dose.
  The incidence of all TEAEs.
Overall Response Rate (ORR) | Every 12 weeks from Day 1 up to 3 years after last dose.
  ORR is the proportion of patients with a confirmed best overall response of complete response (CR) or partial response (PR), as assessed by BICR per RECIST v1.1.
Disease Control Rate (DCR) | Every 12 weeks from Day 1 up to 3 years after last dose.
  DCR is the proportion of patients with a confirmed best overall response of CR, PR, or Stable Disease (SD), as assessed by BICR per RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Marpadga, MD MPH, Study Director — Replimune Inc.
Locations (30):
- United States (29):
  - HonorHealth Research Insisute, Scottsdale, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion(ACP), Aurora, Colorado
  - The Melanoma & Skin Cancer Institute, Englewood, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Mayo Clinic - Jacksonville FL, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt Ingram Cancer Center (Henry-Joyce Cancer Clinic), Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - The University Of Texas Md Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University Of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool, Merseyside, United Kingdom